CLINICAL TRIAL: NCT00708669
Title: A Japanese Prospective, Randomized, Multi-center Trial Comparing the TAXUS Stent and the CYPHER Stent in Patients With Coronary Artery Disease Eligible for PCI.
Brief Title: Japan-Drug Eluting Stents Evaluation; a Randomized Trial
Acronym: J-DESsERT®
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Associations for Establishment of Evidence in Interventions (Other)
Responsible Party: Associations for Establishment of Evidence in Interventions, Associations for Establishment of Evidence in Interventions
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J-DESsERT®, version 1.6
Record Dates: First submitted 2008-06-30; First posted 2008-07-02 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2012-04

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TAXUS group (Active Comparator)
  Interventions: Device: TAXUS stent
- Cypher group (Active Comparator)
  Interventions: Device: Cypher stent

INTERVENTIONS:
Device: TAXUS stent — Compared two kinds of stents:TAXUS stent, approved for commercialization in Japan(March 30th, 2007)
  Arms: TAXUS group
Device: Cypher stent — CYPHER stent, approved for commercialization in Japan(March 25, 2004)
  Arms: Cypher group

SUMMARY:
To evaluate the procedural, short and long term clinical outcomes of the TAXUS stent compared to Cypher stent in coronary arteries of ≥ 2.5 and ≤ 3.75 mm in the reference vessel diameter with a lesion of ≤ 46 mm (by visual observation) in routine clinical settings in Japan.

DETAILED DESCRIPTION:
In these days, meta-analyses have been conducted in large scale and small scale studies, but there has been no conclusion yet stating which one of the stents, either Cypher stent or TAXUS stent, is superior to the other. In specific disease condition such as in diabetic patients, it has been reported that Paclitaxel (TAXUS stent) is more suitable than Sirolimus (Cypher stent), due to the difference in the action mechanisms of the drugs. Since TAXUS stent was recently approved in Japan, we decided to conduct a randomized multi-center comparative study to compare Cypher stent and TAXUS stent regarding the clinical endpoint (target vessel failure for 8 months). The study is powered to show equivalence between the 2 stents in all patients, and to show superiority of the TAXUS stent in the diabetic patient population. In addition, for selected patients, quantitative coronary angiography, intravascular ultrasound, optical coherence tomography, and angioscopy are performed to examine the difference of the two stents more closely.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 20 years old
* Patient suitable for percutaneous coronary intervention (PCI)
* Patient with signed informed consent
* Patient judged suitable to receive anti-platelet drugs (clopidogrel bisulfate or ticlopidine hydrochloride, etc.) in principle for at least 6 months after procedure, and ideally up to 12 months in patients who are not at high risk of bleeding, based on ACC/AHA guideline
* Patient with up to 3 lesions (with ≥ 50% of stenosis) in the maximum of 2 targeted vessels to be treated at once
* Patient with reference vessel diameter (RVD) of 2.5 mm to 3.75 mm by visual observation
* Patient with length of each lesion of up to 46 mm by visual assessment
* Patient eligible for implementation of drug eluting stent.

Exclusion Criteria:

* Patient with any planned treatment in the targeted vessel with a drug eluting stent other than in this study
* Patient with acute myocardial infarction (AMI) (including non-ST segment elevation MI) developed within 7 days before the procedure
* Patient participating in a currently ongoing registry or clinical study, or receiving a treatment which may affect the endpoints of this study
* Patient of childbearing potential with a positive pregnancy test within 14 days before the procedure, or lactating
* Patient who has history of allergy against Sirolimus, Paclitaxel, polymers or stainless steel
* Patient who has history of side-effect against anti-platelet drugs or anti-coagulation drugs
* Patient with serious hepatic dysfunction
* Patient with left ventriculogram ejection fraction of 35% or less
* Patient with three target vessels in need of PCI treatment
* Patient with serious renal dysfunction (serum creatinine value 2mg/dL or higher)
* Patient currently receiving artificial dialysis
* Patient with a malignant tumor (cancer) diagnosed within 5 years before the procedure
* Patient who has received PCI treatment within the past one year
* Patient with chronic total occlusion (CTO) or TIMI flow 2 or less
* Patient with >50% stenosis in left main coronary artery
* Patient with >50% stenosis in side branch ostial for which stenting in the side branch lesion is required (KBT for side branch is accepted)
* Patient with in-stent restenosis in the target lesion implanted with a bare-metal or drug eluting stent
* Patient who has target lesion in saphenous vein graft
* Patient judged non-eligible by the physician in charge.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3500 (Estimated)
Dates: Start 2008-03; Primary Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Target Vessel Failure (TVF) at 8 months post-procedure(assessed prior to routine angiography) in Overall study population | 8 months

SECONDARY OUTCOMES:
Target Vessel Failure (TVF) at 8 months post-procedure (assessed prior to routine angiography) in diabetic group | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Shinsuke Nanto, M.D, Study Chair — Non-profit organization(NPO); "Associations for Establishment of Evidence in Intervations"
Locations (122):
- Japan (122):
  - Aichi Medical University Hospital, Aichi
  - Japan Labour Health and Welfare Organization, Kansai Rosai Hospital, Amagasaki
  - Asahikawa-Kosei General Hospital, Asahikawa
  - Sakakibara Memorial Hospital, Fuchū
  - Fukui Cardiovascular Center, Fukui
  - Fukuoka University Hospital, Fukuoka
  - Gifu Prefectural General Medical Center, Gifu
  - Seirei Hamamatsu General Hospital, Hamamatsu
  - Hekinan Municipal Hospital, Hekinan
  - Saitama Medical University International Medical Center, Hidaka
  - Koto Memorial Hospital, Higashiōmi
  - Kansai Medical University Hirakata Hospital, Hirakata
  - Hiratsuka Kyosai Hospital, Hiratsuka
  - Hirosaki University School of Medicine and Hospital, Hirosaki
  - Hiroshima University Hospital, Hiroshima
  - Tsuchiya General Hospital, Hiroshima
  - Iizuka Hospital, Iizuka
  - Saiseikai Imabari Hospital, Imabari
  - Nippon Medical School Chiba Hokusoh Hospital, Inzai
  - Iwaki Kyoritsu Hospital, Iwaki
  - Rinku General Medical Center, Izumisano
  - Juntendo University Shizuoka Hospital, Izunokuni
  - Setsunan General Hospital, Kadoma
  - Ishikawa Prefectural Central Hospital, Kanazawa
  - Kanazawa Cardiovascular Hospital, Kanazawa
  - Nara Medical University Hospital, Kashihara
  - Japan Labour Health and Welfare Organization, Kanto Rosai Hospital, Kawasaki
  - Kawasaki Saiwai Hospital, Kawasaki
  - Kagawa University Hospital, Kida
  - Kimitsu Chuo Hospital, Kisarazu
  - Kokura Memorial Hospital, Kitakyushu
  - Kobe University Hospital, Kobe
  - Chikamori Hospital, Kochi
  - Hoshi General Hospital, Kōriyama
  - Kumamoto Chuo Hospital, Kumamoto
  - Saiseikai Kumamoto Hospital, Kumamoto
  - Kawasaki Medical School Hospital, Kurashiki
  - Kurume University Hospital, Kurume
  - St.Mary's Hospital, Kurume
  - Japanese Red Cross Kyoto Daini Hospital, Kyoto
  - Koseikai Takeda Hospital, Kyoto
  - Kyoto-Katsura Hospital, Kyoto
  - Mie Heart Center, Mie
  - Miki City Hospital, Miki
  - Miyazaki Medical Association Hospital, Miyazaki
  - Memorial Heart Center Iwate Medical University, Morioka
  - Shiga Medical Center for Adults, Moriyama
  - Musashino Red Cross Hospital, Musashino
  - Tachikawa General Hospital, Nagaoka
  - Kouseikai Hospital, Nagasaki
  - Nagoya daiichi red cross Hospital, Nagoya
  - Nagoya Daini Red Cross Hospital, Nagoya
  - Nagoya Memorial Hospital, Nagoya
  - Okayama Red Cross General Hospital, Okayama
  - Okayama University Hospital, Okayama
  - Sakakibara Heart Institute of Okayama, Okayama
  - National Hospital Organization Osaka National Hospital, Osaka
  - Osaka City University Hospital, Osaka
  - Osaka General Medical Center, Osaka
  - Osaka Police Hospital, Osaka
  - Ogaki Municipal Hospital, Ōgaki
  - Oita Cardiovascular Hospital, Ōita
  - OitaOka Hospital, Ōita
  - Omihachiman Community Medical Center, Ōmihachiman
  - Kitasato University Hospital, Sagamihara
  - Iwatsuki-minami Hospital, Saitama
  - Japan Labour Health and Welfare Organization, Osaka Rosai Hospital, Sakai
  - Caress Sapporo Hokko Memorial Hospital, Sapporo
  - Caress Sapporo Tokeidai Hospital, Sapporo
  - Hokkaido Social Insurance Hospital, Sapporo
  - Sapporo Orthopaedic Cardio-vascular Hospital, Sapporo
  - Teine Keijinkai Hospital, Sapporo
  - Sendai Kousei Hospital, Sendai
  - Sendai Open Hospital, Sendai
  - Tohoku Koseinenkin Hospital, Sendai
  - Jichi Medical University Hospital, Shimotsuke
  - National Cerebral and Cardiovascular Center, Suita
  - Osaka University Graduate School of Medicine, Suita
  - Kagawa Prefectural Central Hospital, Takamatsu
  - Ayase Heart Hospital, Tokyo
  - Edogawa Hospital, Tokyo
  - Itabashi Chuo Medical Center, Tokyo
  - Jikei University Hospital, Tokyo
  - Juntendo University Hospital, Tokyo
  - Juntendo University Nerima Hospital, Tokyo
  - Kanto Medical Center NTT EC, Tokyo
  - Keio University Hospital, Tokyo
  - Mitsui Memorial Hospital, Tokyo
  - Nihon University School of Medicine Itabashi Hospital, Tokyo
  - Nippon Medical School Hospital, Tokyo
  - Showa University Hospital, Tokyo
  - St. Luke's International Hospital, Tokyo
  - Teikyo University Hospital, Tokyo
  - The Cardiovascular Institute Hospital, Tokyo
  - Toho University Ohashi Medical Center, Tokyo
  - Toho University Omori Medical Center, Tokyo
  - Tokyo Medical University Hospital, Tokyo
  - Tokyo Metropolitan Hiroo Hospital, Tokyo
  - Tokyo Women's Medical University Hospital, Tokyo
  - Toranomon Hospital, Tokyo
  - Tomishiro Central Hospital, Tomishiro
  - Toyama Prefectural Central Hospital, Toyama
  - Toyama Red Cross Hospital, Toyama
  - Fujita Health University Hospital, Toyoake
  - Toyohashi Heart Center, Toyohashi
  - Tsuchiura Kyodo Hospital, Tsuchiura
  - Tsuyama Central Hospital, Tsuyama
  - Uwajima City Hospital, Uwajima
  - Wakayama Medical University Hospital, Wakayama
  - Yamagata Prefectural Central Hospital, Yamagata
  - Saiseikai Yamaguchi Hospital, Yamaguchi
  - Japan Labour Health and Welfare Organization, Kumamoto Rosai hospital, Yatsushiro
  - Japan Labour Health and Welfare Organization, Yokohama Rosai Hospital, Yokohama
  - Kanagawa Cardiovascular and Respiratory Center, Yokohama
  - Kikuna Memorial Hospital, Yokohama
  - Saiseikai Yokohamashi Tobu Hospital, Yokohama
  - Showa University Fujigaoka Hospital, Yokohama
  - Showa University Northern Yokohama Hospital, Yokohama
  - Yokohama City University General Medical Center, Yokohama
  - Yokohama Sakae Kyosai Hospital, Yokohama
  - Yokosuka General Hospital Uwamachi, Yokosuka
  - Tottori University Hospital, Yonago